CLINICAL TRIAL: NCT02829216
Title: Functional Profiling of the Hematopoietic Stem Cell Niche in Graft Versus Host Disease Mediated Bone Marrow Insufficiency
Brief Title: Graft-versus-host Disease Associated Myelosuppression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: Bone marrow GvHD
Record Dates: First submitted 2016-05-17; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Abnormal Hematopoiesis; Allogenic Disease; Graft vs Host Disease
Keywords: myelosuppression; mesenchymal stromal cells
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to measure the frequency, functionality and phenotype of bone marrow-derived mesenchymal stromal cells in patients after allogeneic hematopoietic stem cell transplantation. Furthermore, the immune cell infiltrate of the bone marrow will be monitored at the same time. These results will be correlated with the extent of cytopenia and clinical graft-versus-host disease grading.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* acute myeloid leukemia
* myelodysplastic syndrome
* hematopoietic stem cell transplantation

Exclusion Criteria:

* not willing to take part

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AML/MDS receiving an allogeneic hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Changes in the amount of mesenchymal stromal cells after allogeneic hematopoietic stem cell transplantation | up to 1 year after allogeneic hematopoietic stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Malte von Bonin, MD, Principal Investigator — Medizinische Klinik und Poliklinik I, Universitätsklinikum, TU Dresden
Locations (1):
- Medizinische Klinik und Poliklinik I, Universitätsklinikum, TU Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No